CLINICAL TRIAL: NCT03331094
Title: Adult Scoliosis Correction by Bipolar Mini-invasive Assembly Without Graft
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: SCOSANGREFF
Record Dates: First submitted 2017-10-24; First posted 2017-11-06 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Scoliosis
MeSH Terms: conditions — Scoliosis | interventions — Surgical Procedures, Operative; Transplantation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- surgery with graft: The procedure is to place a metal instrumentation (rods and screws) in contact with the spine to correct the deformity. Added to this is a graft between the vertebrae that will allow a bone bridge of ankylosis making the spine completely rigid.
  Interventions: Procedure: Surgery with graft
- surgery without graft: Adult scoliosis surgery is performed with instrumentation without grafting: the teams use variable stiffness rods made of metal or PEEK.
  Interventions: Procedure: surgery without graft

INTERVENTIONS:
Procedure: Surgery with graft — arthrodesis with autologous bone graft and using pedicular ilio-sacred EUROS ® screw
  Groups: surgery with graft
Procedure: surgery without graft — arthrodesis without bone graft using pedicular ilio-sacred EUROS ® screw
  Groups: surgery without graft

SUMMARY:
The objective of the study will be to estimate the correction obtained with a metallic instrumentation, by mini-invasive technique with bipolar assembly and ilio-sacred EUROS ®) screw , without transplant at the adult as compared to that obtained with the surgery with complete exhibition of the rachis and bone graft.

ELIGIBILITY:
Inclusion Criteria:

* age >18
* under guardianship
* vertebral deformation >20°
* accept to participate

Exclusion Criteria:

* minor patient
* surgery not including the pelvis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: every patient with a scoliosis responding to the criteria above recovering for surgery
Sampling Method: Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2016-12-06 (Actual); Primary Completion 2023-11-15 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
change of Cobb angle | change from baseline Cobb angle at 6 months
  Cobb angle represent the degree of curvature of the scoliosis

CONTACTS AND LOCATIONS:
Overall Officials: WOLFF Stephane, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France